CLINICAL TRIAL: NCT05088694
Title: The Optimization and Evaluation of the Extremism and Intolerance Curriculum for the Kingdom of Bahrain.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Jeffrey Milroy, Assistant Professor, University of North Carolina, Greensboro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-FY21-66
Record Dates: First submitted 2021-09-13; First posted 2021-10-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Norm, Social; Literacy; Resistance Skills; Beliefs About Consequences; Decision Making Skills; Empathy; Tolerance; Open Mindedness; Active Citizenship; Anti-extremism
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Classrooms assigned to the intervention group will receive the Peaceful Coexistence (middle school) or Anti-extremism (high school) curricula.
  Interventions: Behavioral: Peaceful Coexistence
- No intervention (No Intervention): Classrooms assigned to the No intervention group will receive general information during their sessions.

INTERVENTIONS:
Behavioral: Peaceful Coexistence — The Peaceful Coexistence intervention seeks to target important risk and protective factors related to tolerance and acceptance.
  The Anti-Extremism intervention seeks to take the same risk and protective factors covered in the Peaceful Coexistence intervention and have students' psychosocial factors shift their skills and behavior.
  Other Names: Anti-Extremism
  Arms: Intervention

SUMMARY:
Researcher from UNC Greensboro have partnered with Prevention Strategies and key stakeholders from the Kingdom of Bahrain to conduct a study using the innovative, engineering-inspired methodological approach, the Multiphase Optimization Strategy (MOST), to optimize and evaluate the Peaceful Coexistence and Anti-Extremism middle and high school curricula. No other curriculum targeting tolerance and/or extremism has been optimized using the state-of-the-art MOST methodology. The overall goal of the project is that the optimized versions of Peaceful Coexistence and Anti-Extremism curricula will be used across the Kingdom of Bahrain and translated for use in other countries to combat the spread of extremism and intolerance. Additionally, the D.A.R.E. keepin' it REAL (kiR) and D.A.R.E. myPlaybook high school programs will be evaluated as part of the Peaceful Coexistence and Anti-Extremism evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Public or private Bahraini middle or high school students.
* In addition to the main evaluation questions, the following groups will also be included to make programmatic improvements.
* Parents of above mentioned middle or high school students.
* D.A.R.E. Officers teaching middle school and high school D.A.R.E. in Bahrain.

Exclusion Criteria:

* None

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Norms about intolerance | immediately post intervention
  Participant's mean rating of norms related to intolerance of others measured by the intolerance norms scale.
Dignity | immediately post intervention
  Mean rating of dignity reported by participants measured by the Jacelon Attributed Dignity Scale.
Plurality | immediately post intervention
  Mean rating of religious plurality reported by participants using the Religious Plurality scale.
Beliefs about consequences | immediately post intervention
  Mean rating of participant beliefs about consequences related to not listening to different opinions of others measured by the Beliefs about intolerance consequences scale.
Source literacy | immediately post intervention
  Mean rating of participants' reported source literacy measured by the Source literacy scale.
Resistance skills | immediately post intervention
  Mean rating of participants' reported efficacy to resist religiously, politically, or socially extreme sentiments measured by the Resistance skills scale.
Decision making | immediately post intervention
  Mean rating of participants' report of decision making skills measured by the Decision making skills scale.
Empathy | immediately post intervention
  Mean rating of participants' empathy toward people and opinions that are different from their own measured by the Emotional Quotient Scale.
Tolerance of different opinions and behaviors of others | immediately post intervention
  Mean rating pf participants' reporting of expectations of others based on tolerant behaviors measured by the Tolerance of others scale.
Open Mindedness to differing opinions | immediately post intervention
  Mean ratings of participants' report of open mindedness of differing political, social, and religious ideals measured by the Open Minded Cognition Scale.
Non-Violent Conflict Resolution | immediately post intervention
  Mean rating of participants' ideals related to non-violent conflict resolution measured by the Normative Beliefs about Aggression Scale.
Community values | immediately post intervention
  Mean rating of participants' opinions related to their expectations of other as it pertains to extremist behaviors measured by the community values scale.

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Greensboro, Greensboro, North Carolina, United States